CLINICAL TRIAL: NCT01457417
Title: A Two Part Phase 1 Multicenter Open-label Study of DKN-01 Given Intravenously. Part A: Dose-Escalation in Patients With Multiple Myeloma or Advanced Solid Tumors. Part B: Expansion Cohort in Patients With Relapsed / Refractory Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of DKN-01 in Multiple Myeloma or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100; DEK-DKK1-P100 (Other: Healthcare Pharmaceuticals); LY2812176 (Other: Healthcare Pharmaceuticals)
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma; Solid Tumors; Non-Small Cell Lung Cancer
Keywords: Cancer; Oncology
MeSH Terms: conditions — Multiple Myeloma; Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 75 milligram (mg) DKN-01 Part A (Experimental): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle.
  PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
  Interventions: Drug: DKN-01
- 150 mg DKN-01 Part A (Experimental): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle.
  PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
  Interventions: Drug: DKN-01
- 300 mg DKN-01 Part A (Experimental): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle.
  PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
  Interventions: Drug: DKN-01
- 600 mg DKN-01 Part A (Experimental): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle.
  PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
  Interventions: Drug: DKN-01
- 300 mg DKN-01 Part B (Experimental): Dose Confirmation: Once the MTD had been established or the highest planned dose level completed, 300 mg of DKN-01 was administered as IV on days 1 and 15 of every 28 day cycle.
  Interventions: Drug: DKN-01

INTERVENTIONS:
Drug: DKN-01 — DKN-01 will be administered intravenously (IV) once a week over 30 minutes (min) and 2 hours (max) for 75, 150 and 300 mg. At 600 mg, DKN-01 will be administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: 3 participants will be treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation will occur sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching maximum tolerated dose (MTD) are met (or highest planned dose study group is completed). Cycle 1 will define the dose limiting toxicity (DLT) that governs dose escalation. PART B - Dose Confirmation: Once the MTD is established (or the highest planned dose level), 300 mg of DKN-01 will be administered IV on days 1 and 15 of every 28 day cycle.
  Other Names: Formerly LY2812176

SUMMARY:
The purpose of this trial is to characterize the safety and toxicity of DKN-01 by determining a maximum-tolerated dose and associated dose limiting toxicity. To evaluate the pharmacodynamic response in patients with cancer. To characterize the pharmacokinetic parameters of DKN-01 in cancer patients who are intolerant to standard/approved therapies.

DETAILED DESCRIPTION:
Part A of this trial consists of 4 treatment arms of DKN-01. It is a dose escalation study in patients with multiple myeloma or advanced solid tumors. Patients must be refractory or intolerant to all standard/approved therapy(ies). At each dose level, 3 subjects will be treated. If none of the 3 subjects develop a dose limiting toxicity after a minimum of 4 weeks of treatment, subsequent dose escalation will proceed according to the same schedule. Part B consists of dose confirmation in patients with NSCLC. Patients must be refractory or intolerant to all standard/approved therapy(ies). Approximately 15 patients may be enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

Part A: Patients with histological or cytological confirmed multiple myeloma or advanced solid tumors. For multiple myeloma, must have symptomatic myeloma as defined by the International Myeloma Working Group inclusive of measurable serum and/or urine monoclonal protein (M-protein) or for those without elevations they must have measurable increased concentrations of free light chains

Part B: Patients with previously treated, histologically confirmed advanced NSCLC with progressive disease requiring therapy

Parts A and B:

* Refractory or intolerant to all standard/approved therapy(ies)
* Patients with solid tumors must have one or more metastatic tumors measurable on computed tomography (CT) scan using Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Radiation for symptomatic lesions outside the central nervous system (CNS) must have been completed at least 2 week prior to study enrollment
* Treated brain metastases will be allowed, if they are asymptomatic. Patients must be off corticosteroids for at least 2 week prior to study entry
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1
* Life expectancy of at least 3 months
* Ambulatory patients greater than or equal to (≥) 30 years of age
* Females with child bearing potential must have a negative serum pregnancy test within 7 days of study entry
* Acceptable liver function, renal function, hematologic status
* Urinalysis - No clinically significant abnormalities
* Acceptable coagulation status:

  * Prothrombin Time/Partial Thromboplastin Time (PT/PTT) ≤ 1.2 x upper limit of normal (ULN) (unless receiving anticoagulation therapy - eligibility based upon INR)
  * International Normalization Ratio (INR) ≤ 1.6 (unless receiving anticoagulant therapy)

    * Receiving warfarin; INR ≤ 3.0 and no active bleeding
* For men and women of child-producing potential, the use of effective contraceptive methods during the study and for women 18 months following the last dose of study drug
* Available for the study duration and willing to follow procedures
* Serum calcium:

  * Solid tumors only: within normal limits
  * Multiple myeloma: ≤ 11.5 milligrams per deciliter (mg/dL)

Exclusion Criteria:

* History of osteonecrosis of the hip or evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan considered clinically significant or may impact the interpretation of the scan. Degenerative changes of the hip joint are not exclusionary
* Unable to tolerate the confinement/noise of an MRI scanner or have any contraindication for MRI
* New York Heart Association Class 3 or 4, cardiac disease, myocardial infarction, unstable arrhythmia, or evidence of ischemia
* Have Fridericia-corrected QT interval (QTcF) > 470 millisecond (msec) (female) or > 450 (male), or history of congenital long QT syndrome.
* Active, uncontrolled bacterial, viral, or fungal infections
* Pregnant or nursing women
* Radiation therapy, surgery, or chemotherapy, within 1 month prior to study entry
* Previously treated with an anti-Dickkopf-related protein 1 (DKK-1) therapy
* Significant allergy to a biological pharmaceutical therapy
* History of major organ transplant
* Had an autologous or allogenic bone marrow transplant, current acute leukemia, colon, prostate, breast or small cell lung cancer, osteoblastic lesions, concomitant disease known to influence calcium metabolism including hyperparathyroidism, hyperthyroidism and/or Paget's disease of bone
* Unwillingness / inability to comply with procedures
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Serious nonmalignant disease
* Receiving other investigational agent or have received other investigational agent within last 30 days or 5 half-lives, whichever is longer
* Receiving lithium chloride (LiCl)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndi Sirard, MD, Study Director — Heatlhcare Pharmaceuticals
Locations (8):
- United States (8):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - New York Oncology Hematology, P.C., Albany, New York
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Texas Oncology - Baylor, Charles A. Sammonds Cancer Center, Dallas, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associated, Norfolk, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight sites in the United States participated in the study and 7 of them enrolled patients. The Date of First Enrollment was 16 Jan 2012, and the Date of Last Completed was 06 Dec 2013.
Pre-assignment Details: Part A enrolled patients with histologically or cytologically confirmed multiple myeloma or advanced solid tumors. A dose escalation procedure was followed. Part B enrolled patients with non-small cell lung cancer. Following screening (up to 28 days prior to first treatment) if entry criterion was met, patients were eligible for enrollment.
Groups:
- 75 Milligram (mg) DKN-01 Part A (QW); 600 mg DKN-01 Part A (Q2W): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
- 150 mg DKN-01 Part A (QW): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method will be guided by the incidence of DLTs during the first cycle.
- 300 mg DKN-01 Part A (QW): DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) was met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
- 300 mg DKN-01 Part B (Q2W): Dose Confirmation: Once the MTD had been established or the highest planned dose level completed, 300 mg of DKN-01 was administered as IV on days 1 and 15 of every 28 day cycle.
Period: Overall Study
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Started | 3 | 3 | 4 | 3 | 19
Completed | 3 | 3 | 4 | 3 | 19
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 150 mg DKN-01 Part A: DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) were met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method will be guided by the incidence of DLTs during the first cycle.
- 300 mg DKN-01 Part A: DKN-01: DKN-01 was administered intravenously (IV) once a week over a minimum of 30 minutes and up to a maximum of 2 hours for dose levels of 75 mg, 150 mg and 300 mg. At the 600 mg dose level, DKN-01 was administered by IV on days 1 and 15 of each cycle. PART A - Dose Escalation: Study group of 3 participants were treated with a 28 day cycle of DKN-01 at an assigned dose level until disease progression. Dose escalation occurred sequentially over the doses of 75, 150, 300, and 600 mg until the criteria for reaching the maximum tolerated dose (MTD) was met or the highest planned dose study group was completed. Cycle 1 defined the dose limiting toxicity (DLT) period that governs dose escalation. The dose escalation method was guided by the incidence of DLTs during the first cycle.
- Total: Total of all reporting groups
Arm/Group | 75 Milligram (mg) DKN-01 Part A | 150 mg DKN-01 Part A | 300 mg DKN-01 Part A | 600 mg DKN-01 Part A | 300 mg DKN-01 Part B | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 19 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.77) | 66.3 (8.62) | 65.0 (19.20) | 68.3 (8.96) | 65.4 (9.25) | 65.0 (10.29)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 2 | 1 | 10 | 17
  >=65 years | 0 | 2 | 2 | 2 | 9 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 1 | 9 | 18
  Male | 2 | 0 | 0 | 2 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Summary of Total Adverse Events (AE)
Description: Total Adverse Events (AE), total treatment emergent adverse events (TEAE), total Serious Adverse Events (SAE), and total dose-limiting toxicity (DLT) for both Parts A and B.
Time Frame: Baseline to study completion (approximately 3 months)
Population: Safety analyses were based on the full analysis set (FAS), which was defined as all patients who received at least one dose of study treatment during Part A or Part B of the study.
Measure: Number; unit: Events
Groups:
- Total: Total across all treatment groups
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 19 | 32
Events
  Total AEs | 39 | 58 | 35 | 11 | 87 | 230
  Total TEAEs | 39 | 58 | 35 | 9 | 87 | 228
  Total SAEs | 2 | 7 | 3 | 0 | 11 | 23
  Total DLTs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Summary of Patients With Adverse Events (AE)
Description: Number of patients who had Adverse Events (AE) including treatment related treatment emergent adverse events (TEAE), Common Toxicity Criteria for Adverse Effects (CTCAE), and Serious Adverse Events (SAE) for both Parts A and B. Severity was coded to NCI CTCAE version 4.02. For maximum severity and relationship, patients were counted only once in the most severe or most related category.
Time Frame: Baseline to study completion (approximately 3 months)
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 19 | 32
Patients
  At Least One AE | 3 | 3 | 4 | 3 | 16 | 29
  At Least One TEAE | 3 | 3 | 4 | 3 | 16 | 29
  At Least One SAE | 1 | 2 | 1 | 0 | 7 | 11
  Retracted SAE | 1 | 2 | 0 | 0 | 2 | 5
  SAE related to study drug | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Maximum CTCAE - Grade 1 Mild | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Maximum CTCAE - Grade 2 Moderate | 2 | 1 | 1 | 3 | 6 | 13
  TEAE of Maximum CTCAE - Grade 3 Severe | 0 | 2 | 3 | 0 | 9 | 14
  TEAE of Maximum CTCAE - Grade 4 Life Threatening | 1 | 0 | 0 | 0 | 0 | 1
  TEAE of Maximum CTCAE - Grade 5 Death | 0 | 0 | 0 | 0 | 1 | 1
  TEAE Grade ≥ 3 assessed as study drug related | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Maximum Relationship - Related | 1 | 2 | 3 | 1 | 8 | 15
  TEAE of Maximum Relationship - Not Related | 2 | 1 | 1 | 2 | 8 | 14
  At Least One TEAE Leading to Drug Withdrawal | 0 | 1 | 0 | 0 | 3 | 4
  At Least One TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  At Least One TEAE with Outcome of Death | 0 | 0 | 0 | 0 | 1 | 1

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration - Time Curve (AUC) of DKN-01
Description: Area under the DKN-01 serum concentration-time profile curve during the dosing interval (AUC0-tau) after the first and fourth infusion for both Parts A and B. Cycle 1 Day 1 included once per week (QW) dosing groups and every two weeks (Q2W) dosing groups.
Time Frame: Cycle 1 Day 1 (first dose, all groups)
Population: All patients who received at least one dose of study treatment during Part A or Part B of the study.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 18
hr*ng/mL | 1942552.08830 (780226.768012) | 4381685.27190 (402701.016054) | 10860453.92050 (2319628.494223) | 18103276.11133 (1250736.327819) | 18398867.35928 (5107540.116369)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration - Time Curve (AUC) of DKN-01
Description: Area under the DKN-01 serum concentration-time profile curve during the dosing interval (AUC0-tau) after the first and fourth infusion for both Parts A and B. Cycle 1 day 22 included only QW dosing groups.
Time Frame: Cycle 1 Day 22 (Fourth Dose for QW)
Population: All patients who received at least one dose of study treatment during Part A study.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
hr*ng/mL | 5663382.27007 (3919446.471337) | 15815320.60770 (5614032.150398) | 25639949.52467 (4567585.003954) |  |

5. Secondary Outcome: Pharmacokinetic: Maximum Plasma Concentration (Cmax) of DKN-01
Description: Peak DKN-01 serum concentration (Cmax) after the first and fourth infusion on Cycle 1 Weeks 1 and 4, for both Parts A and B. Cycle 1 Day 1 included once per week (QW) dosing groups and every two weeks (Q2W) dosing groups.
Time Frame: Cycle 1 Day 1 (first dose, all groups)
Population: All patients who received at least one dose of study treatment during Part A or Part B of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 18
ng/mL | 22756.09897 (7665.992335) | 47838.87113 (4193.154016) | 130105.94600 (25705.162094) | 183063.33233 (34635.447386) | 119837.93546 (43565.776017)

6. Secondary Outcome: Pharmacokinetic: Maximum Plasma Concentration (Cmax) of DKN-01
Description: Peak DKN-01 serum concentration (Cmax) after the fourth infusion on Cycle 1 Weeks 1 and 4, for both Parts A and B. Cycle 1 day 22 included only QW dosing groups.
Time Frame: Cycle 1 Day 22 (Fourth dose for QW groups)
Population: All patients who received at least one dose of study treatment during Part A of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
ng/mL | 43203.11520 (25085.681036) | 105148.29720 (29480.395189) | 224382.14533 (28438.209780) |  |

7. Secondary Outcome: Progression Free Survival (PFS) in Patients Who Are Refractory or Intolerant to Standard/Approved Therapies
Description: For both Parts A and B. PFS was defined as the time from the date of signed informed consent to the first date of objectively determined progressive disease (Progression is defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and International Multiple Myeloma Working Group (IMWG)) or death from any cause. For patients who were still alive at the time of analysis (i.e, data cut-off date) and without evidence of tumor progression, PFS was censored at the date of the most recent objective progression-free observation.
Time Frame: Time from the date of signed informed consent to the first date of objectively determined progressive disease or death from any cause
Population: All patients who received at least one dose of study treatment during Part A or Part B of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 19
Months | 3.4 [2.2 to 4.7] | 2.4 [1.7 to 3.3] | 2.1 [1.5 to 2.2] | 2.1 [2.1 to 2.2] | 2.2 [1.5 to 2.9]

8. Secondary Outcome: Overall Survival (OS) in Patients With Relapsed or Refractory NSCLC
Description: For Part B only. OS was defined as the time from the date of signed informed consent to the date of death from any cause. For patients who were still alive as of the data cut-off date, OS time was censored on the date of the patient's last contact (last contact for patients in post-discontinuation was the last date of contact in long-term follow-up eCRF).
Time Frame: Time from the date of signed informed consent to the date of death from any cause
Population: For patients who are still alive as of the data cut-off date, OS time will be censored on the date of the patient's last contact (last contact for patients in post-discontinuation = last Date of Contact in Long Term Follow-up eCRF).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 19
Months | 6.6 [4.1 to 10.1]

9. Secondary Outcome: Objective Response Rate (ORR) in Oncologic Patients Who Are Refractory or Intolerant to Standard/Approved Therapies
Description: For both Parts A and B. Objective response rate is defined as the number of patients with overall best response of complete response (CR) or partial response (PR)
Time Frame: Part A: Every 2 months; Part B: after 1 month and every two cycles thereafter
Population: All patients with NSCLC who received at least one dose of study treatment during Part A or Part B of the study. One Patients from the 300 mg QW treatment group, and two patients from 300 mg Q2W treatment group did not have assessments performed after Baseline.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 17
Participants | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 60.2] | 0 [0 to 70.8] | 1 [.1 to 26.0]

10. Secondary Outcome: Objective Response Rate (ORR) in Patients With Relapsed or Refractory Non-small Cell Lung Cancer (NSCLC)
Description: FAS : For both Parts A and B. Objective response rate is defined as the number of patients with overall best response of complete response (CR) or partial response (PR)
Time Frame: Part A: Every 2 months; Part B: after 1 month and every two cycles thereafter
Population: FAS : NSCLC - All patients with NSCLC who received at least one dose of study treatment during Part A or Part B of the study. Two patients in treatment group 300 mg Q2W did not have assessments performed after Baseline.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 75 Milligram (mg) DKN-01 Part A (QW) | 150 mg DKN-01 Part A (QW) | 300 mg DKN-01 Part A (QW) | 600 mg DKN-01 Part A (Q2W) | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 2 | 1 | 0 | 2 | 17
participants | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] |  | 0 [0.0 to 84.2] | 1 [0.1 to 26.0]

11. Primary Outcome: Progression Free Survival (PFS) in Patients With Relapsed or Refractory Non-small Cell Lung Cancer (NSCLC)
Description: For Part B only. The distribution of PFS was estimated using the Kaplan-Meier (KM) method. PFS was defined as the time from the date of signed informed consent to the first date of objectively determined progressive disease (Progression is defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and International Multiple Myeloma Working Group (IMWG)) or death from any cause. For patients who were still alive at the time of analysis (ie, data cut-off date) and without evidence of tumor progression, PFS was censored at the date of the most recent objective progression-free observation.
Time Frame: as for outcome 7
Population: Patients with advanced NSCLC receiving the study drug at 300 mg every 2 weeks in Part B
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 300 mg DKN-01 Part B (Q2W)
Number analyzed (Participants) | 18
months | 2.2 [1.5 to 2.9]

ADVERSE EVENTS:
Time Frame: Entirety of the study. 1 year, 3 months.
Description: Safety analyses were based on the full analysis set (FAS), which was defined as all patients who received at least one dose of study treatment during Part A or Part B of the study. Assessments up to 30 days after the date of last dose of study medication (for serious adverse events and unresolved study drug-related AEs) were included.
Arm/Group | 75 Milligram (mg) DKN-01 Part A | 150 mg DKN-01 Part A | 300 mg DKN-01 Part A | 600 mg DKN-01 Part A | 300 mg DKN-01 Part B
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/4 | 0/3 | 6/19
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 75 Milligram (mg) DKN-01 Part A (N=3) | 150 mg DKN-01 Part A (N=3) | 300 mg DKN-01 Part A (N=4) | 600 mg DKN-01 Part A (N=3) | 300 mg DKN-01 Part B (N=19)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN MANAGEMENT (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 Milligram (mg) DKN-01 Part A (N=3) | 150 mg DKN-01 Part A (N=3) | 300 mg DKN-01 Part A (N=4) | 600 mg DKN-01 Part A (N=3) | 300 mg DKN-01 Part B (N=19)
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 4
FATIGUE (General disorders) | 0 | 2 | 3 | 0 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 6
VOMITTING (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 2
ASTHENIA (General disorders) | 1 | 1 | 1 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results shall not be made before the publication by Sponsor. If there is no multi-site publication within 18 months after the Study completion/termination at all sites, the Site shall have the right to publish its results. Prior to submitting to public release the Sponsor has 60 days from receipt to review and comment. The Site shall, upon Sponsor's request, further delay publication/presentation for up to 120 days to allow Sponsor to protect its interests.